CLINICAL TRIAL: NCT04786327
Title: Intrabony Defects Management Using Growth Factor Enhanced Matrix Versus Platelet Rich Fibrin Utilizing Minimally Invasive Surgical Technique. A Randomized Clinical and Radiographic Trial.
Brief Title: Minimally Invasive Flap With Platelet Rich Fibrin or Growth Factor Enhanced Matrix in Treatment of Intrabony Defect
Acronym: RCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, malak mohamed shoukheba, associate prof, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2021-02-25; First posted 2021-03-08 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Periodontal Regeneration
Keywords: Chronic periodontitis; Intra-bony defects; Minimally invasive surgical technique; Platelet rich fibrin,; Growth factor enhanced matrix 21S
MeSH Terms: conditions — Chronic Periodontitis | interventions — Edetic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- treated by using Minimally invasive flap only. (Placebo Comparator): 7 sites treated with Minimally invasive flap only
  Interventions: Procedure: Minimal invasive flap technique
- Minimally invasive flap with root conditioning (EDTA) and platelet rich fibrin . (Experimental): 7 sites treated with Minimally invasive flap plus EDTA root conditioning and application of platelet rich fibrin graft
  Interventions: Procedure: Minimally invasive flap with root conditioning (EDTA) and platelet rich fibrin
- MIST with root conditioning (EDTA) and GEM 21S . (Experimental): 7 sites treated with Minimally invasive flap plus EDTA root conditioning and application of growth factor enhanced matrix GEM21S
  Interventions: Combination Product: minimally invasive flap with root contioning by EDTA and growth factor enhanced matrix GEM21S

INTERVENTIONS:
Procedure: Minimal invasive flap technique — contained defect treated with Minimally invasive flap
  Other Names: regenerative surgery
  Arms: treated by using Minimally invasive flap only.
Procedure: Minimally invasive flap with root conditioning (EDTA) and platelet rich fibrin — contained defect treated by Minimally invasive flap with root conditioning (EDTA) and platelet rich fibrin graft
  Other Names: regenerative surgery
  Arms: Minimally invasive flap with root conditioning (EDTA) and platelet rich fibrin .
Combination Product: minimally invasive flap with root contioning by EDTA and growth factor enhanced matrix GEM21S — contained defect treated with Minimally invasive flap with root conditioning (EDTA) and growth factor enhanced matrix application in the defect
  Other Names: regenerative surgery
  Arms: MIST with root conditioning (EDTA) and GEM 21S .

SUMMARY:
Twenty-one intra-bony defects in fifteen systemically healthy patients with moderate to severe chronic periodontitis were randomly classified into 3 groups, 7 sites each. Group І treated by MIST alone, group ІІ treated by MIST + ethylenediamine-tetraaceticacid (EDTA) + PRF and group III treated by MIST + EDTA + GEM 21S. The clinical parameters including probing pocket depth (PPD), clinical attachment level (CAL) and bleeding on probing (BOP), were recorded at baseline, 3, 6 and 9 months post-surgery. Cone beam computed tomography (CBCT) was performed at baseline and 9 months post-surgery to evaluate bone level and bone density

DETAILED DESCRIPTION:
: Twenty-one intra-bony defects in fifteen systemically healthy patients with moderate to severe chronic periodontitis were randomly classified into 3 groups, 7 sites each. Group І treated by MIST alone, group ІІ treated by MIST + ethylenediamine-tetraaceticacid (EDTA) + PRF and group III treated by MIST + EDTA + GEM 21S. The clinical parameters including probing pocket depth (PPD), clinical attachment level (CAL) and bleeding on probing (BOP), were recorded at baseline, 3, 6 and 9 months post-surgery. Cone beam computed tomography (CBCT) was performed at baseline and 9 months post-surgery to evaluate bone level and bone density.

ELIGIBILITY:
Inclusion Criteria:

• Presence of at least one tooth with PPD and CAL loss of ≥ 5 mm associated with an intra-bony defect of ≥ 2 mm according to Cortellini and Tonetti, 2007

Exclusion Criteria:

* Patients with uncontrolled or poorly controlled diabetes, life-threatening conditions, or requiring antibiotic prophylaxis were excluded.
* Smokers
* Pregnant patients.
* Patients with aggressive periodontitis.
* Patients with multiple interconnected vertical defect walls.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
the change in probing pocket depth | 9 months
  the change in probing pocket depth was measured at baseline, 3,6 and 9 months evaluation period using periodontal probe
the change bleeding on probing score | 9 months
  the change in bleeding on probing measured at baseline,3,6 and 9 months evaluation period
the change Clinical attachment level | 9 months
  the change in Clinical attachment level measured at baseline, 3,6 and 9 months using the periodontal probe
Cone beam radiograph | 9 months
  Cone beam radiograph for measuring the change in area of the defect, depth of the depth and bone density at baseline, 3, 6 and 9 month post operative treatment using OnDemand software of cone beam

CONTACTS AND LOCATIONS:
Overall Officials: malak m shoukheba, phd, Principal Investigator — tanta university faculty of dentistry
Locations (1):
- Malak Mohamed Shoukheba, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No